CLINICAL TRIAL: NCT02189265
Title: Assessing the Impact of Smoke-free Legislation on Perinatal Health in the Netherlands
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: Maastricht University Medical Center (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); The Netherlands Perinatal Registry (PRN) (Unknown)
Responsible Party: Principal Investigator, Jasper Been, Dr., University of Edinburgh
Other Study IDs: TRF NR-0166-1.3
Record Dates: First submitted 2014-07-03; First posted 2014-07-14 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Premature Birth; Perinatal Mortality; Infant, Low Birth Weight; Stillbirth; Infant Mortality; Sudden Infant Death; Infant, Very Low Birth Weight; Infant, Small for Gestational Age
Keywords: Live birth [MeSH]; Infant [MeSH]; Infant, newborn [MeSH]; Second-hand smoke; Tobacco smoke pollution [MeSH]; Smoke-free; Smoke-free policy [MeSH]
MeSH Terms: conditions — Premature Birth; Perinatal Death; Stillbirth; Infant Death; Sudden Infant Death

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Biospecimen Retention: None Retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Full cohort: All singleton births in the Netherlands. Stillbirths are excluded from the denominator for all outcomes other than perinatal mortality, stillbirth and congenital anomalies.
  Interventions: Other: Smoke-free legislation

INTERVENTIONS:
Other: Smoke-free legislation — The intervention under study is the ban on smoking in workplaces, and in bars and restaurants implemented in the Netherlands on January 1st, 2004 and July 1st, 2008, respectively.

SUMMARY:
The purpose of this study is to investigate whether there has been a change in perinatal outcomes following the phased smoking ban introduction (January 2004 for workplaces; July 2008 for bars and restaurants) workplaces in the Netherlands.

DETAILED DESCRIPTION:
Primary research questions

1. Is the phased introduction of smoke-free legislation in The Netherlands associated with reductions in adverse perinatal outcomes (e.g. perinatal mortality, preterm birth, small for gestational age)?
2. How do these associations compare with those described for other European countries in comparable studies (i.e. Belgium (Cox 2013), England (Been et al under review), Scotland (Mackay 2012))?

Study design Retrospective cohort study (using prospective routinely collected health care data)

Study population All singleton births in the Netherlands between January 1st 2000 and December 31st 2011.

Intervention The intervention under study is the ban on smoking in workplaces, and in bars and restaurants implemented in the Netherlands on January 1st, 2004 and July 1st, 2008, respectively.

Inclusion and exclusion criteria We will include all registered singleton births in the Netherlands occurring between January 1st, 2000 and December 31st, 2011. This is the maximum time period surrounding the ban's introduction for which the required birth data are available through the data source. Multiple pregnancies, neonates with chromosomal anomalies, pregnancies with unknown gestational age, pregnancies that ended before 24 weeks and pregnancies resulting in the birth of a child weighing less than 500 grams will be excluded.

Outcome

The primary outcomes are:

* Perinatal mortality (stillbirth + early neonatal mortality, i.e. within the first 7 days of life)
* Preterm birth (live birth with gestational age <37+0 weeks)
* Small for gestational age (SGA; live birth with birth weight below 10th centile; The Dutch PRN reference curves for birth weight by gestational age according to parity, sex and ethnic background will be used)

To assess whether smoke-free legislation had a selective impact on certain subgroups of outcomes we furthermore identified a number of secondary outcomes:

* Stillbirth (born dead from 24+0 weeks of gestation)
* Early neonatal mortality (live birth and death within first 7 days)
* Very preterm birth (live birth with gestational age <32+0 weeks)
* Low birth weight (live birth with birth weight <2500 grams)
* Very low birth weight (live birth with birth weight <1500 grams)
* Very small for gestational age (live birth with birth weight below percentile 2.3rd centile)
* Major congenital anomalies (based on reported associations with antenatal smoke exposure (Hackshaw 2011)).

Data sources Individual level health care data will be extracted from The Netherlands Perinatal Registry (PRN). Linked midwifery, obstetric, and neonatal data are available from 2000 to 2011 (including 2011).

Data extraction and handling All relevant variables regarding our outcomes, as well as relevant potential confounders will be extracted from the database.

Sample size Power calculation for interrupted time series modelling is complicated given the complexity of the analysis. Similar previous studies have demonstrated statistically significant and clinically relevant effects of smoke-free legislation on preterm birth (Cox 2013; Mackay 2012; Page 2012), low birth weight (Mackay 2012), SGA (Mackay 2012; Kabir 2013), and perinatal mortality (Mackay et al. and Been et al. both under review). Given the larger population size of the Netherlands as opposed to the regions in which these studies were carried out (except for Been et al. under review), we expect our study to have sufficient power to detect similar effect sizes, should these be present.

Statistical analysis Incidences for each outcome will be presented graphically for each time period to facilitate visualisation of temporal fluctuations and trends in changes of incidence levels. To facilitate timing of the events, date of delivery and expected term date are required for each pregnancy. Data will be presented as outlined in different Tables. Interrupted time series analyses with adjustment for potential confounders will be performed to assess the associations between implementation of smoke-free legislation and primary and secondary outcome measures. Individual-level analysis will be performed using logistic regression analysis. The models will account for the underlying temporal trend in incidence, and will allow for a sudden change in incidence ('step change') following the introduction of the smoking bans. We will test and adjust for any non-linearity in the underlying time trends, and seasonality will be accounted as appropriate.

Sensitivity analyses (primary outcomes only) In recent years, gestational age is usually estimated based on early ultrasonography findings, which is more reliable than estimation based on the last menstrual period. Although the method of ascertainment is not recorded in PRN, there is an item indicating 'certainty' of the gestational age, which is positive in about 93% of records. For the primary outcomes preterm birth and SGA we will perform a sensitivity analysis including only cases in whom gestational age estimation is considered reliable according to this item.

Recent perinatal management changes have been implemented in The Netherlands resulting in increased active management of babies born at the edge of viability (i.e. 23-24 weeks gestation) (NVOG 2010). This has resulted in increased survival at this gestational age as well as altered management of 25-26 week infants, which likely affects the number of babies born preterm (although this effect is expected to be small given the small percentage of all preterm babies being born at this stage), as well as mortality indicators. For the primary outcomes preterm birth and perinatal mortality we will therefore perform a sensitivity analysis excluding babies born before 26 completed weeks of gestation.

Smoking during pregnancy is known to be underreported in the PRN database. Definitions between different caregivers differ; (any) smoking and heavy smoking (>20 cigarettes daily). We will consider performing subgroup analyses of the impact of smoke-free legislation on the primary outcomes according to maternal smoking status during pregnancy.

In a sensitivity analysis we will investigate whether smoke-free legislation has any differential impact on spontaneous preterm birth versus medically indicated preterm birth.

All analyses will be performed using Stata 13.0.

ELIGIBILITY:
Data are obtained via The Netherlands Perinatal Registry (PRN) (6). All registered stillbirths and livebirths occurring in the Netherlands between 1 January 2000 and 31 December 2011 are included.

Inclusion Criteria:

* Singleton birth occurring in the Netherlands between January 1st, 2000 and December 31st, 2011
* Liveborn (for all outcomes other than stillbirth and congenital anomalies)

Exclusion Criteria:

* No chromosomal anomalies

Max Age: 1 Week | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All singleton births in the Netherlands. Stillbirths are excluded from the denominator for all outcomes other than stillbirths and congenital anomalies.
Sampling Method: Probability Sample
Enrollment: 2069695 (Actual)
Dates: Start 2000-01; Primary Completion 2011-12 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Perinatal mortality | from 24+0 weeks gestation (for stillbirth); up to 7 days postnatally (for early neonatal mortality)
  stillbirth (i.e. intrauterine death from 24+0 weeks gestation) or early neonatal mortality (i.e. death within the first 7 days postnatally)
Preterm birth | gestational age >= 24+0 weeks and <37+0 weeks
  live birth with gestational age >= 24+0 weeks and <37+0 weeks
Small for gestational age | gestational age >= 24+0 weeks
  live birth at gestational age >= 24+0 weeks with birth weight below 10th centile

SECONDARY OUTCOMES:
Stillbirth | gestational age >= 24+0 weeks
  born dead from 24+0 weeks of gestation
Early neonatal mortality | up to 7 days postnatally after live birth at gestational age >= 24+0 weeks
  death within first 7 days after live birth at gestational age >= 24+0 weeks
Very preterm birth | gestational age >= 24+0 weeks and <32+0 weeks
  live birth with gestational age >= 24+0 weeks and <32+0 weeks
Low birth weight | gestational age >= 24+0 weeks
  live birth at gestational age >= 24+0 weeks with birth weight <2500 grams
Very low birth weight | gestational age >= 24+0 weeks
  live birth at gestational age >= 24+0 weeks with birth weight <1500 grams
Very small for gestational age | gestational age >= 24+0 weeks
  live birth at gestational age >= 24+0 weeks with birth weight below 2.3rd centile
Major congenital anomalies | gestational age >= 24+0 weeks
  birth at >= 24+0 weeks of gestation with a major birth defect (birth defects known to be influenced by antenatal smoke exposure based on recent systematic review (Hackshaw 2011))

CONTACTS AND LOCATIONS:
Overall Officials: Jasper V Been, MD MPH PhD, Principal Investigator — Allergy and Respiratory Research Group, Centre for Population Health Sciences, The University of Edinburgh, Edinburgh, UK
Locations (2):
- Academic Medical Centre, Amsterdam, North Holland, Netherlands
- Centre for Population Health Sciences, The University of Edinburgh, Edinburgh, Midlothian, United Kingdom

REFERENCES:
- [Background] Cox B, Martens E, Nemery B, Vangronsveld J, Nawrot TS. Impact of a stepwise introduction of smoke-free legislation on the rate of preterm births: analysis of routinely collected birth data. BMJ. 2013 Feb 14;346:f441. doi: 10.1136/bmj.f441. PMID 23412829
- [Background] Mackay DF, Nelson SM, Haw SJ, Pell JP. Impact of Scotland's smoke-free legislation on pregnancy complications: retrospective cohort study. PLoS Med. 2012;9(3):e1001175. doi: 10.1371/journal.pmed.1001175. Epub 2012 Mar 6. PMID 22412353
- [Background] Page RL 2nd, Slejko JF, Libby AM. A citywide smoking ban reduced maternal smoking and risk for preterm births: a Colorado natural experiment. J Womens Health (Larchmt). 2012 Jun;21(6):621-7. doi: 10.1089/jwh.2011.3305. Epub 2012 Mar 8. PMID 22401497
- [Background] Kabir Z, Daly S, Clarke V, Keogan S, Clancy L. Smoking ban and small-for-gestational age births in Ireland. PLoS One. 2013;8(3):e57441. doi: 10.1371/journal.pone.0057441. Epub 2013 Mar 26. PMID 23555561
- [Background] Hackshaw A, Rodeck C, Boniface S. Maternal smoking in pregnancy and birth defects: a systematic review based on 173 687 malformed cases and 11.7 million controls. Hum Reprod Update. 2011 Sep-Oct;17(5):589-604. doi: 10.1093/humupd/dmr022. Epub 2011 Jul 11. PMID 21747128
- [Background] de Laat MW, Wiegerinck MM, Walther FJ, Boluyt N, Mol BW, van der Post JA, van Lith JM, Offringa M; Nederlandse Vereniging voor Kindergeneeskunde; Nederlandse Vereniging voor Obstetrie en Gynaecologie. [Practice guideline 'Perinatal management of extremely preterm delivery']. Ned Tijdschr Geneeskd. 2010;154:A2701. Dutch. PMID 21429260
- [Derived] Peelen MJ, Sheikh A, Kok M, Hajenius P, Zimmermann LJ, Kramer BW, Hukkelhoven CW, Reiss IK, Mol BW, Been JV. [Tobacco control policies and perinatal health]. Ned Tijdschr Geneeskd. 2017;161:D563. Dutch. PMID 28120730
- [Derived] Peelen MJ, Sheikh A, Kok M, Hajenius P, Zimmermann LJ, Kramer BW, Hukkelhoven CW, Reiss IK, Mol BW, Been JV. Tobacco control policies and perinatal health: a national quasi-experimental study. Sci Rep. 2016 Apr 22;6:23907. doi: 10.1038/srep23907. PMID 27103591